CLINICAL TRIAL: NCT07073235
Title: Neuroplastic Changes and Effects of Intermittent Theta Burst Stimulation (iTBS) on Motor Recovery of Upper and Lower Extremity in Chronic Stroke Patients
Brief Title: Effects of Intermittent Theta Burst Stimulation (iTBS) on Motor Recovery of Lower Extremity in Chronic Stroke Patients
Acronym: NIMBLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Danderyd Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Susanne Palmcrantz, PhD, Associate Professor, Reg Physiotherapist, Danderyd Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: iTBS-study lower extremity
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Hemiparesis After Stroke; Chronic Stroke Patients; Hemiplegia; Ambulatory Difficulty
Keywords: stroke; iTBS; TMS; Trancranial Magnetic Stimulation; Cerebellum; Chronic stroke patients; Balance; Walking; Hemiparesis; intermittent Theta Burst Stimulation
MeSH Terms: conditions — Stroke; Hemiplegia; Mobility Limitation; Paresis

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Contralesional cerebellum iTBS and conventional rehabilitation (Experimental): The experimental group will receive intermittent theta burst stimulation on the contralesional cerebellum followed by 45 minutes of conventional rehabilitation interventions involving the lower extremity led or instructed by a physiotherapist.
  Interventions: Device: Intermittent Theta Burst Stimulation
- Contralesional cerebellum sham-iTBS and conventional rehabilitation (Sham Comparator): The placebo group will get sham intermittent theta burst stimulation on the contralesional cerebellum followed by 45 minutes of conventional rehabilitation interventions involving the lower extremity led or instructed by a physiotherapist.
  Interventions: Device: Sham Intermittent Theta Burst Stimulation

INTERVENTIONS:
Device: Intermittent Theta Burst Stimulation — iTBS protocol: 600 pulses at 80% of AMT for 190 sec on the contralesional cerebellum, targeted with the support of a neuronavigational system, 15 sessions over a period of 5 weeks
  Other Names: iTBS; TMS
  Arms: Contralesional cerebellum iTBS and conventional rehabilitation
Device: Sham Intermittent Theta Burst Stimulation — It is identical to its active version, replicates operational sounds, and delivers a very shallow magnetic field to mimic the sensation of magnetic stimulation.
  Arms: Contralesional cerebellum sham-iTBS and conventional rehabilitation

SUMMARY:
This study aims to evaluate the effects and clinical feasibility of non-invasive brain stimulation protocols, specifically intermittent Theta Burst Stimulation, as part of rehabilitation interventions for motor recovery of lower extremity in the chronic phase after stroke.

It also seeks to explore the underlying mechanisms by investigating changes of functional and structural brain networks.

DETAILED DESCRIPTION:
In this randomized control trial (RCT) group A will receive iTBS while group B will receive sham iTBS. Both groups will directly after the intervention receive 45 minutes of conventional physical therapy 3 times per week for 5 weeks, a total of 15 interventions by a blinded physiotherapist. For the iTBS intervention a Magstim Rapid² stimulator will be used also equipped with a Cadwell Sierra Summit EMG system [for motor evoked potential (MEP) measurements] and an ANT Visor2™ neuronavigation system [for navigated transcranial magnetic stimulation (TMS) interventions]. The iTBS parameters that will be used are: 600 pulses under 190 seconds at 80 % of Active Motor Threshold (AMT). The contralesional cerebellum will be targeted. The participants and clinical assessors will be blinded to the intervention.

All the patients will undergo advanced neuroimaging examinations before and after the intervention period. The exams will be then compared to identify neuroplastic changes in brain circuits.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Chronic stroke (>6 months)
* Residual hemiparesis FAC ≥3

Exclusion Criteria:

* Metal implants
* Epilepsy/seizures
* Pregnancy
* Claustrophobia (related to MRIs exams)
* Severe cognitive impairment
* Untreated or unstable depression/anxiety
* Other disabilities prohibiting intensive physical training

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
miniBest test | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  measures dynamic balance, functional mobility, and gait. It is a 14-item test scored on a 3-level ordinal scale. The score ranges from 0 to 28 points. A higher score indicates better balance.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment - Lower Extremity | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  used to quantify sensorimotor function recovery after a stroke. It is a 43 item test scored on a 3-level ordinal scale. The score ranges from 0 to 86 points. A higher score indicates higher sensorimotor recovery.
Modified Ashworth Scale (MAS) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  Assesses spasticity on a 6 point scale/muscle (0p no impairment, 5p max impairment/muscle).
Neuroflexor | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  Medical technology device. Assesses spasticity by identifying the neural, viscous and elastic components during passive movement using a biomechanical algorithm (presented in Newton)
Lower Extremity Motor Coordination Test (LEMOCOT) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  assesses motor coordination deficits after stroke. The LEMOCOT assesses how many times a participant can alternately touch a proximal and distal target with their big toe within 20 seconds. Higher scores indicate better motor coordination in the lower extremity.
6 minutes walk test | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  assess submaximal aerobic/functional walking capacity, community walking prediction. Assesses walking endurance in meters walked. Longer distances indicate better walking capacity.
Functional Ambulation Categories (FAC) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  evaluates ambulation ability. It ranges from 0 to 5. Higher score indicates more independent ambulation.
Falls Efficacy Scale Swedish version (FES-S) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  measure the level of concern about falling during social and physical activities inside and outside home. The total score ranges from 0 to 130. A higher total score on the FES-S indicates greater confidence in performing the activities without falling.
Walking impact scale (MSWS-12 S) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  Assesses self-perceived limitations in walking. The score ranges from 12 to 60 (12p no impairments, 60p max impairment).
Canadian Occupational Performance Measure | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  Captures the participant´s perception of performance in everyday living, over time and is used to set and evaluate goals of an intervention
Montreal Cognitive Assessment (MoCA) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  Assesses mental function (0p max impairment summed up to 30p no detected impairment)
Stroke Impact Scale (SIS) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  is a self-report questionnaire that evaluates disability and health-related quality of life after stroke. It has 8 domains: strength, hand function, mobility, physical and instrumental activities of daily living (ADL and IADL), memory and thinking, communication, emotion, and social participation. It uses a 5-point Likert scale to assess the difficulty of performing various tasks within each domain. Higher scores indicate better outcome
Motor Evoked Potentials (MEPs) | At baseline, after completion of the 5 week intervention to assess change as well at 12 weeks follow up.
  electrical signals recorded from neural tissue or muscle following activation of central motor pathways. MEPs assess the integrity of descending motor pathways.
Resting state functional MRI (rs-fMRI) | At baseline and after completion of the 5 week intervention to assess changes.
  a method aimed at examining intrinsic networks in the brain while no task is performed (rest); this is to estimate correlations between brain regions.
Diffusion Tensor Imaging (DTI) | At baseline and after completion of the 5 week intervention to assess changes
  a method aimed at mapping structural correlations between brain regions.

OTHER OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | At baseline.
  quantifies stroke severity based on weighted evaluation findings. The total NIHSS score ranges from 0 to 42, with higher scores indicating more severe strokes, categorized as follows: minor stroke (1-4), moderate stroke (5-15), moderate to severe stroke (16-20), and severe stroke (21-42).
Barthel Index (BI) | At baseline.
  measures a person's ability to complete activities of daily living (ADL). Scores range from 0 to 100, categorized as follows: Total dependence (0-20), Severe dependence (21-60), Moderate dependence (61-90), Slight dependence (91-99), and Independence (100).
Theoretical Framework of Acceptability questionnaire | After completion of the 5 week intervention to assess acceptability.
  to assess the acceptability of healthcare interventions, based on the developed Theoretical Framework of Acceptability (TFA). It uses a 5-point Likert scale to assess acceptability of the intervention. Higher scores indicate higher acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Palmcrantz, PhD, Associate Professor, Principal Investigator — Dep of Clinical Sciences, Karolinska Institutet
Locations (1):
- Department of Rehabilitation Medicine, Danderyd Hospital, Danderyd, Stockholm 18288, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramnani N. The primate cortico-cerebellar system: anatomy and function. Nat Rev Neurosci. 2006 Jul;7(7):511-22. doi: 10.1038/nrn1953. PMID 16791141
- [Background] Wang J, Wu Z, Hong S, Ye H, Zhang Y, Lin Q, Chen Z, Zheng L, Qin J. Cerebellar transcranial magnetic stimulation for improving balance capacity and activity of daily living in stroke patients: a systematic review and meta-analysis. BMC Neurol. 2024 Jun 15;24(1):205. doi: 10.1186/s12883-024-03720-1. PMID 38879485
- [Background] Wang C, Zhang Q, Zhang L, Zhao D, Xu Y, Liu Z, Wu C, Wu S, Yong M, Wu L. Comparative efficacy of different repetitive transcranial magnetic stimulation protocols for lower extremity motor function in stroke patients: a network meta-analysis. Front Neurosci. 2024 Feb 15;18:1352212. doi: 10.3389/fnins.2024.1352212. eCollection 2024. PMID 38426021
- [Background] Koch G, Bonni S, Casula EP, Iosa M, Paolucci S, Pellicciari MC, Cinnera AM, Ponzo V, Maiella M, Picazio S, Sallustio F, Caltagirone C. Effect of Cerebellar Stimulation on Gait and Balance Recovery in Patients With Hemiparetic Stroke: A Randomized Clinical Trial. JAMA Neurol. 2019 Feb 1;76(2):170-178. doi: 10.1001/jamaneurol.2018.3639. PMID 30476999
- [Background] Jiang T, Wei X, Wang M, Xu J, Xia N, Lu M. Theta burst stimulation: what role does it play in stroke rehabilitation? A systematic review of the existing evidence. BMC Neurol. 2024 Feb 1;24(1):52. doi: 10.1186/s12883-023-03492-0. PMID 38297193
- [Background] Fan H, Song Y, Cen X, Yu P, Biro I, Gu Y. The Effect of Repetitive Transcranial Magnetic Stimulation on Lower-Limb Motor Ability in Stroke Patients: A Systematic Review. Front Hum Neurosci. 2021 Sep 1;15:620573. doi: 10.3389/fnhum.2021.620573. eCollection 2021. PMID 34539362
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Christiansen MG, Senko AW, Anikeeva P. Magnetic Strategies for Nervous System Control. Annu Rev Neurosci. 2019 Jul 8;42:271-293. doi: 10.1146/annurev-neuro-070918-050241. Epub 2019 Apr 2. PMID 30939100
- [Background] Qi S, Tian M, Rao Y, Sun C, Li X, Qiao J, Huang ZG. Applying transcranial magnetic stimulation to rehabilitation of poststroke lower extremity function and an improvement: Individual-target TMS. Wiley Interdiscip Rev Cogn Sci. 2023 Mar;14(2):e1636. doi: 10.1002/wcs.1636. Epub 2022 Nov 27. PMID 36437474
- [Background] Fan J, Fu H, Xie X, Zhong D, Li Y, Liu X, Zhang H, Zhang J, Huang J, Li J, Jin R, Zheng Z. The effectiveness and safety of repetitive transcranial magnetic stimulation on spasticity after upper motor neuron injury: A systematic review and meta-analysis. Front Neural Circuits. 2022 Nov 8;16:973561. doi: 10.3389/fncir.2022.973561. eCollection 2022. PMID 36426136